CLINICAL TRIAL: NCT02124291
Title: Effect of Assisted Hatching on Vitrified Embryo Transfer Clinical Outcome
Acronym: VitHatSZMC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient enrollment
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Principal Investigator, Volodarsky-Perel Alexander, MD, MD, Shaare Zedek Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VitHatSZMC
Record Dates: First submitted 2014-04-23; First posted 2014-04-28 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2017-04

CONDITIONS: Complications Associated With Artificial Fertilization; Placenta; Implantation; Pregnancy
Keywords: In Vitro Fertilization; Vitrification; Frozen Embryo; Assisted Hatching; Pregnancy Rate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- No Assisted Hatching (No Intervention): No Assisted Hatching
- Assisted Hatching (Active Comparator): Mechanical Assisted Hatching - artificial rupture of the embryo external glycoprotein layer (Zona Pellucida) before embryo transfer.
  Interventions: Device: Mechanical Assisted Hatching

INTERVENTIONS:
Device: Mechanical Assisted Hatching — The technique of assisted hatching using partial zona pellucida dissection to create an artificial opening of the zona pellucida of early cleaved embryos. While the embryo is stabilized by a holding pipette of micromanipulator, the zona pellucida is pierced with a microneedle that is pushed tangentially through the space between the zona pellucida and blastomeres until it pierces through the zona pellucida again.
  Arms: Assisted Hatching

SUMMARY:
The objective of study is to assess the possible impact of assisted hatching on the implantation, pregnancy rate and delivery rate after transfer of vitrified-warmed human embryos.

DETAILED DESCRIPTION:
The embryo implantation rate in assisted reproduction procedures is 20%, which leads to a low clinical pregnancy rate (35%), and even lower live birth rate (25%), per cycle started. Low embryo quality, poor endometrial receptivity, difficulties during the blastocyst hatching process are frequently denoted as the main reasons for the low implantation rate in humans.

The artificial rupture or thinning of the zona pellucida before embryo transfer-assisted hatching (AH)-has been proposed to foster spontaneous hatching and improve embryo implantation rates. Despite great effort, the clinical relevance of AH remains controversial and elusive.

There is a great importance of AH during frozen embryo cycles. Due to previous studies there is no precise answer about the value of AH performed on cryopreserved-thawed embryos. As far as is known, there is no clinical data to indicate the effects of AH on vitrified-warmed embryo transfer.

The objective of this prospective study is to assess the possible impact of assisted hatching on the implantation, pregnancy rate and delivery rate after transfer of vitrified-warmed human embryos.

Eligibility criteria: women age 18-42, cleavage-stage embryo transfer, less than seven IVF cycles with fresh embryo transfer, high quality embryos.

Procedure: mechanical Assisted Hatching

Primary Outcome: delivery rate Secondary Outcome: implantation rate, pregnancy rate and delivery rate.

ELIGIBILITY:
Inclusion Criteria:

* women age 18-42,
* cleavage-stage embryo transfer,
* less than seven IVF cycles with fresh embryo transfer,
* high quality embryos.

Exclusion Criteria:

* out of 18-42 y.o.
* blastocyst embryo transfer
* more or equal to seven IVF cycles with fresh embryo transfer
* low quality embryos

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2014-06; Primary Completion 2015-12 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
delivery rate | 9 months

SECONDARY OUTCOMES:
implantation rate | 1 month
clinical pregnancy rate | 2 months

OTHER OUTCOMES:
multifetal pregnancy | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Volodarsky-Perel, MD, Principal Investigator — Shaare Zedek Medical Center, Jerusalem, Israel.; Avi Tsafrir, MD, Study Chair — Shaare Zedek Medical Center, Jerusalem, Israel
Locations (1):
- Shaare Zedek Medical Center, Jerusalem, Israel

REFERENCES:
- [Background] Sagoskin AW, Levy MJ, Tucker MJ, Richter KS, Widra EA. Laser assisted hatching in good prognosis patients undergoing in vitro fertilization-embryo transfer: a randomized controlled trial. Fertil Steril. 2007 Feb;87(2):283-7. doi: 10.1016/j.fertnstert.2006.07.1498. Epub 2006 Nov 13. PMID 17094975
- [Background] Fang C, Li T, Miao BY, Zhuang GL, Zhou C. Mechanically expanding the zona pellucida of human frozen thawed embryos: a new method of assisted hatching. Fertil Steril. 2010 Sep;94(4):1302-1307. doi: 10.1016/j.fertnstert.2009.08.014. Epub 2009 Sep 26. PMID 19782973
- [Background] Valojerdi MR, Eftekhari-Yazdi P, Karimian L, Ashtiani SK. Effect of laser zona pellucida opening on clinical outcome of assisted reproduction technology in patients with advanced female age, recurrent implantation failure, or frozen-thawed embryos. Fertil Steril. 2008 Jul;90(1):84-91. doi: 10.1016/j.fertnstert.2007.06.005. Epub 2007 Sep 24. PMID 17889864
- [Background] Ng EH, Naveed F, Lau EY, Yeung WS, Chan CC, Tang OS, Ho PC. A randomized double-blind controlled study of the efficacy of laser-assisted hatching on implantation and pregnancy rates of frozen-thawed embryo transfer at the cleavage stage. Hum Reprod. 2005 Apr;20(4):979-85. doi: 10.1093/humrep/deh724. Epub 2005 Jan 21. PMID 15665025
- [Background] Martins WP, Rocha IA, Ferriani RA, Nastri CO. Assisted hatching of human embryos: a systematic review and meta-analysis of randomized controlled trials. Hum Reprod Update. 2011 Jul-Aug;17(4):438-53. doi: 10.1093/humupd/dmr012. Epub 2011 Apr 7. PMID 21474527
- [Background] Valojerdi MR, Eftekhari-Yazdi P, Karimian L, Hassani F, Movaghar B. Effect of laser zona thinning on vitrified-warmed embryo transfer at the cleavage stage: a prospective, randomized study. Reprod Biomed Online. 2010 Feb;20(2):234-42. doi: 10.1016/j.rbmo.2009.11.002. Epub 2009 Nov 18. PMID 20113961
- [Background] Carney SK, Das S, Blake D, Farquhar C, Seif MM, Nelson L. Assisted hatching on assisted conception (in vitro fertilisation (IVF) and intracytoplasmic sperm injection (ICSI). Cochrane Database Syst Rev. 2012 Dec 12;12(12):CD001894. doi: 10.1002/14651858.CD001894.pub5. PMID 23235584
- [Background] Gabrielsen A, Agerholm I, Toft B, Hald F, Petersen K, Aagaard J, Feldinger B, Lindenberg S, Fedder J. Assisted hatching improves implantation rates on cryopreserved-thawed embryos. A randomized prospective study. Hum Reprod. 2004 Oct;19(10):2258-62. doi: 10.1093/humrep/deh434. Epub 2004 Aug 19. PMID 15319388
- [Background] Wan CY, Song C, Diao LH, Li GG, Bao ZJ, Hu XD, Zhang HZ, Zeng Y. Laser-assisted hatching improves clinical outcomes of vitrified-warmed blastocysts developed from low-grade cleavage-stage embryos: a prospective randomized study. Reprod Biomed Online. 2014 May;28(5):582-9. doi: 10.1016/j.rbmo.2014.01.006. Epub 2014 Jan 27. PMID 24631166